CLINICAL TRIAL: NCT04199000
Title: Clinical and Basic Investigations Into Congenital Disorders of Glycosylation
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Seattle Children's Hospital (Other); Children's Hospital of Philadelphia (Other); University of Pittsburgh (Other); Boston Children's Hospital (Other); Tulane University School of Medicine (Other); Baylor College of Medicine (Other); University of Minnesota (Other); Children's Hospital Colorado (Other); Sanford-Burnham Medical Research Institute (Other); University of Utah (Other); University of Alabama at Birmingham (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eva Morava-Kozicz, Principal Investigator, Icahn School of Medicine at Mount Sinai
Other Study IDs: Mayo 19-005187; U54NS115198-01 (NIH)
Record Dates: First submitted 2019-12-08; First posted 2019-12-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Congenital Disorders of Glycosylation
Keywords: CDG; CDDG; Congenital Disorders of Glycosylation; Congenital Disorders of Deglycosylation; ALG1; ALG3; ALG6; ALG12; ALG13; COG6; DPAGT1; DPM1; EDEM3; MAN1B1; MPDU1; MPI; NGLY1; PGAP3; PGM1; PIGA; PIGG; PIGN; PIGS; PIGT; PMM2; SLC35A2; SLC35C1; SLC39A8; SRD5A3; SSR4; FUT8; GALNT2; MAN2B2; VMA21
MeSH Terms: conditions — Congenital Disorders of Glycosylation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Stool, urine, and blood can be retained for biomarker testing. DNA may be a part of this testing in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to study the natural history of congenital disorders of glycosylation and its causes and treatments.

DETAILED DESCRIPTION:
The investigators are conducting a natural history study of patients with congenital disorders of glycosylation (CDG). The study will look into the progression of the disease amongst the participants and also look at the clinical symptoms and how they vary amongst different diseased population groups. The participants will be asked to fill out questionnaires either on their own or with a provider that will grade the severity of disease and document symptoms and diet. Participants will have an opportunity to submit blood, urine, and stool samples that will be tested for biomarkers for CDG.

Participants will also complete dietary food records, physical exams, CDG scores, and the PROMIS questionnaires to assess disease progression and severity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a genetically, enzymatically, or molecularly confirmed diagnosis of CDG or NGLY1 deficiency

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a genetically, enzymatically, or molecularly confirmed diagnosis of a congenital disorder of glycosylation (CDG) or NGLY1 deficiency, or individuals whose laboratory values are highly suggestive of CDG
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Indicators of Disease Severity and Progression - organ system involvement | Length of study, up to 5 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of the Nijmegen Progression CDG rating scale.
Indicators of Disease Severity and Progression - degree of cognitive disability | Length of study, up to 5 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of the Nijmegen Progression CDG rating scale.
Indicators of Disease Severity and Progression - case-fatality | Length of study, up to 5 years
  Establish the prevalence and severity of specific morbid indicators of disease severity through use of the Nijmegen Progression CDG rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (12):
- United States (12):
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and samples may be shared with other investigators at the discretion of the PI. Only participants who have consented to sharing data/samples will be included in this portion.
Supporting Information: Study Protocol, ICF
Time Frame: Length of study and beyond

REFERENCES:
- See also: Frontiers in Congenital Disorders of Glycosylation (FCDGC) — https://www.rarediseasesnetwork.org/fcdgc